CLINICAL TRIAL: NCT01291823
Title: A Phase II Study of Gefitinib Combined With Radiotherapy in Elderly Patients With Esophageal
Brief Title: Gefitinib Combined With Radiotherapy in Elderly Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: MAO Weimin，XU Yaping, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH10
Record Dates: First submitted 2011-02-04; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Esophageal Cancer
Keywords: gefitinib; radiation; esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Concomitant Gefitinib and radiotherapy (Experimental): Patients received Gefitinib and radiation therapy
  Interventions: Drug: gefitinib; Radiation: Thoracic radiotherapy

INTERVENTIONS:
Drug: gefitinib — gefitinib 250mg/day
Radiation: Thoracic radiotherapy — Thoracic radiotherapy 54-60Gy over 30 fraction

SUMMARY:
Elderly patients with esophageal cancer will receive thoracic radiation therapy 54-60Gy over 30 fractions, and concurrent with Gefitinib.

DETAILED DESCRIPTION:
Purpose: to evaluate the efficacy and toxicity of a concomitant treatment using EGFR-TKI and thoracic radiation in elderly patients with esophageal Cancer.

Methods:Patients(>70 years old) with esophageal Cancer will receive thoracic radiation therapy 54-60 Gy over 30 fractions and concurrent with gefitinib 250mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of esophageal Cancer
* Disease must be encompassed in a radiotherapy field.Patients with celiac, perigastric, mediastinal or supraclavicular adenopathy are eligible
* age:70-85 years
* Written informed consent.
* Performance status of 0 to 2
* Neutrophil count >1.5 x 10 to the 9th power/L and platelets > 100 x 10 to the 9th power/L.
* Hepatic: total bilirubin less than or equal to 1.5 times upper limit of normal (ULN) Alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 2.5 times ULN (or less than or equal to 5 times ULN in case of known liver involvement
* Renal: Serum Creatinine less than or equal to 1.5 times upper limit of normal (ULN)

Exclusion Criteria:

* Evidence of tracheoesophageal fistula, or invasion into the trachea or major bronchi.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
* Prior systemic chemotherapy or radiation therapy for esophageal cancer

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate | 1 month after the thoracic radiotherapy and concurrent gefitinib treatment

SECONDARY OUTCOMES:
The safety (The safety was evaluated according to the National Cancer Institute Common Toxicity Criteria version 3.0.) | 1 month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mao Weimin, MD, Principal Investigator — Zhejiang Cancer Hospital; Xu yaping, MD, Principal Investigator — 0086-571-88122082
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China